CLINICAL TRIAL: NCT03315988
Title: The Effects of an 8-week Vegan Diet on Trimethylamine-N-Oxide (TMAO) Levels and Post-challenge Glucose Levels in Individuals With Dysglycaemia (The Plant Your Health Study)
Brief Title: The Effects of an 8-week Vegan Diet on TMAO Levels and Post-challenge Glucose Levels in Individuals With Dysglycaemia
Acronym: PYH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0625
Record Dates: First submitted 2017-10-04; First posted 2017-10-20 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 2; Heart Diseases
Keywords: type 2 diabetes; vegan diet; TMAO; cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vegan diet (Experimental): Intervention Description and Definition The participants will be asked to follow a diet that excludes foods hypothesised to support the syntheses of TMAO, particularly meat (any), eggs and fish (any). A number of studies suggest that dairy products may also have an effect in modulating TMAO production whereas other studies do not. Therefore, in order to avoid any potential contaminating or confounding effect, dairy products will also be avoided.
  The diet employed in this study is broadly aligned to a vegan diet. The term vegan will be used to aid behaviour change and food choice. For example, an increasing array of products are now pack marked as vegan. The participants will be asked to keep their diet similar to their original and the Registered Dietitian involved in this study will plan their weekly menus accordingly.
  Interventions: Other: Adoption of a vegan diet

INTERVENTIONS:
Other: Adoption of a vegan diet — Adoption of a vegan diet The participants of this study wil be asked to adopt a vegan diet under the supervision of a Registered Dietitian.

SUMMARY:
The amount of people with diabetes mellitus has now reached over 4 million in the United Kingdom. Type 2 diabetes accounts for the majority of all cases of diabetes and increases the risk of many other diseases such as heart problems. Plant based diets are thought to be an effective way to improve markers of health related to type 2 diabetes and heart disease. One way that a plant based diet improves health could be through reducing waste products that are generated in the gut by the bacteria that break down food as part of the digestion process. For example, the digestion of some meats, fish and eggs results in the creation of a substance called Trimethylamine-N-Oxide (TMAO) which has been linked to worse health outcomes in several studies. However, the full impact on TMAO and blood glucose levels of swapping regular meat consumption for a plant based vegan diet is not fully understood and requires further research. Therefore, the aim of this study will be to develop and undertake a clinical trial to investigate the effects of an 8-week vegan diet on TMAO levels and post challenge glucose levels in individuals with dysglycaemia (drug naïve).

The study will be interventional single group prospective trial of adults aged 18-75 years of age from a multi-ethnic population with dysglycaemia (drug naïve). A sample of 29 people will be sought. The dietary intervention (vegan diet) will last 8 weeks. Then, the participants will go back to their normal diet and come for their final visit after a four week follow-up period (week 12). To assess the effectiveness of the intervention, primary and secondary outcome data collected at baseline will be compared with data collected at 1 week, 8 weeks and 12 weeks.

DETAILED DESCRIPTION:
Study Design

Interventional single group prospective trial in a patient population with identified dysglycaemia within the past 36 months defined as 2h post-challenge glucose ≥7.8 mmol/L after a standard oral glucose tolerance test or HbA1c ≥5.7% (39-46 mmol/mol). This phase clinical trial will evaluate the efficacy and underlining mechanisms of a vegan diet in promoting cardiometabolic health in those with dysglycaemia. Specifically, this trial will aim to investigate the effect of an 8-week vegan diet with follow-up at 1, 8 and 12 weeks.

Study Setting

The study will be co-ordinated within the Leicester Biomedical Research Centre (Leicester Diabetes Centre) at the Leicester General Hospital. Clinical measurement sessions will be carried out by the appointed research team. Participants will be asked to visit the study centre on five occasions.

Intervention Description and Definition

The participants will be asked to follow a diet that excludes foods hypothesised to support the syntheses of TMAO, particularly meat (any), eggs and fish (any). A number of studies suggest that dairy products may also have an effect in modulating TMAO production whereas other studies do not. Therefore, in order to avoid any potential contaminating or confounding effect, dairy products will also be avoided.

The diet employed in this study is broadly aligned to a vegan diet. The term vegan will be used to aid behaviour change and food choice. For example, an increasing array of products are now pack marked as vegan. The participants will be asked to keep their diet similar to their original and the Registered Dietitian involved in this study will plan their weekly menus accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* And either:

  * Overweight (White: BMI>25 - <30, South Asian/ Black and minority ethnic group <27.5) with HbA1c between HbA1c ≥5.7% and ≤ 8% (39-64 mmol/mol) identified within the last 36 months
  * Obese: (White: BMI ≥30, South Asian/ Black and minority ethnic group: ≥27.5)
* Male or Female
* Aged 18 - 75 years inclusive
* Able to understand, read and speak the English language to a sufficient level to understand and take part to the study in the investigators opinion
* Have access to a phone, and willing to use it as part of the study
* Regular meat and/or fish eater (at least 3 times per week)-self reported

Exclusion Criteria:

Participant is unwilling or unable to give informed consent

* Non-English speakers
* HbA1c above 8% (64 mmol/mol)
* Taking any form of glucose lowering medication currently or within the last 60 days
* Current smokers
* Current use of vegan or vegetarian diet
* Recent significant weight change (10% or more) over the last 3 months
* Pregnancy/lactation
* Clinical eating disorder as detected by their GP or relevant health professional (e.g. dietitian)
* Have a terminal illness
* Current or recent (within 6 months) oral antibiotics or steroid use as their usage could impact on the gut bacteria profile
* Ongoing CVD (e.g. angina) *

  * In the circumstance that an individual is not sure whether they meet the inclusion/ exclusion criteria, (i.e. they are not sure if they have ongoing CVD) this will be reviewed by a named medic on the delegation of authority log for a clinical decision to be made during baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline TMAO plasma levels at 1, 8 and 12 weeks. | at 1 (+ 5 days) week , 8 (+/- 5 days) weeks and 12 weeks (+/- 5 days)
  urine and plasma samples for TMAO (μM)
Change from Baseline 3-hour post-challenge glucose levels at 1, 8 and 12 weeks. | at 1 (+ 5 days) week , 8 (+/- 5 days) weeks and 12 weeks (+/- 5 days)
  blood samples (mmol/l)

SECONDARY OUTCOMES:
TMAO (μM) urine levels at baseline. | at baseline
  urine samples
Change from Baseline in TMAO urine/plasma levels at 1 week following a vegan diet. | at 1 week (+ 5 days)
  urine and plasma samples; TMAO (μM)
Change from Baseline 3-hour post-challenge glucose levels at 1 week following a vegan diet. | at 1 week (+ 5 days)
  blood samples for glucose (mmol/l)
Change from week 8 in TMAO urine/plasma levels at 4 weeks after diet has returned to normal (week 12). | at 12 weeks (+/- 5 days)
  urine and plasma samples for TMAO (μM)
Change from week 8 in 3-hour post-challenge glucose levels at 4 weeks after diet has returned to normal (week 12). | at 12 weeks (+/- 5 days)
  blood samples for glucose (mmol/l)
Change from Baseline in body composition using dual energy X-ray absorptiometry (DXA) scan at 8 weeks following a vegan diet. | at baseline and week 8 (+/- 5 days)
  DXA Scan
Change from Baseline in biochemical measures of cardiometabolic health including post-challenge insulin at 1 week. | 1 week (+5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including post-challenge insulin at 8 weeks. | 8 weeks (+/- 5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including post-challenge insulin at 12 weeks. | 12 weeks (+/- 5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including fasting lipids and at 1 week. | 1 week (+5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including fasting lipids and inflammatory markers at 8 weeks. | 8 weeks (+/- 5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including fasting lipids at 12 weeks. | 12 weeks (+/- 5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including inflammatory markers at 1 week. | 1 week (+5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including inflammatory markers at 8 weeks. | 8 weeks (+/- 5 days)
  blood samples (mmol/l)
Change from Baseline in biochemical measures of cardiometabolic health including inflammatory markers at 12 weeks. | 12 weeks (+/- 5 days)
  blood samples (mmol/l)
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to body composition. | baseline
  DXA scan
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to body composition. | week 8 (+/- 5 days)
  DXA scan
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to lifestyle factors. | baseline
  3-day diet diaries
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to lifestyle factors. | counselling visit (+5 days)
  3-day diet diaries
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to lifestyle factors. | week 1 (+5 days)
  3-day diet diaries
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to lifestyle factors. | week 8 (+/- 5 days)
  3-day diet diaries
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to lifestyle factors. | week 12 (+/- 5 days)
  3-day diet diaries
The extent to which changes in the primary outcomes are mediated by, or independent of, changes to lifestyle factors. | weeks 1-12
  accelerometers
Semi-structured interviews with the completers, at the end of the study, to investigate perception responses having been on a vegan diet. | at week 12 (+/- 5 days)
  semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Leicester Diabetes Centre, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Argyridou S, Davies MJ, Biddle GJH, Bernieh D, Suzuki T, Dawkins NP, Rowlands AV, Khunti K, Smith AC, Yates T. Evaluation of an 8-Week Vegan Diet on Plasma Trimethylamine-N-Oxide and Postchallenge Glucose in Adults with Dysglycemia or Obesity. J Nutr. 2021 Jul 1;151(7):1844-1853. doi: 10.1093/jn/nxab046. PMID 33784394